CLINICAL TRIAL: NCT00915603
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Weekly Paclitaxel/Bevacizumab +/- Everolimus as First-Line Chemotherapy for Patients With HER2-Negative Metastatic Breast Cancer (MBC)
Brief Title: Trial of Paclitaxel/Bevacizumab +/- Everolimus for Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCRI BRE 154
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Paclitaxel; Bevacizumab; Everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Bevacizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- paclitaxel/bevacizumab/everolimus (Active Comparator): Systemic Therapy
  Interventions: Drug: Everolimus; Drug: Bevacizumab; Drug: Paclitaxel
- paclitaxel/bevacizumab/placebo (Placebo Comparator): Systemic Therapy
  Interventions: Drug: Placebo; Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Everolimus — Everolimus 10mg PO daily continuously for all 28 days of a cycle
  Other Names: Systemic therapy; RAD001; Afinitor
  Arms: paclitaxel/bevacizumab/everolimus
Drug: Bevacizumab — Bevacizumab 10mg/kg IV Days 1 and 15 of 28 day cycle
  Other Names: Systemic therapy; Avastin
  Arms: paclitaxel/bevacizumab/everolimus
Drug: Paclitaxel — Paclitaxel 90mg/m2 1-hour IV infusion Days 1, 8 and 15 of 28 day cycle. Patients will receive standard pre-medication before each paclitaxel treatment to prevent a hypersensitivity reaction.
  Other Names: Systemic therapy; Taxol
  Arms: paclitaxel/bevacizumab/everolimus
Drug: Placebo — Placebo PO daily continuously for all 28 days of a cycle
  Other Names: Systemic therapy
  Arms: paclitaxel/bevacizumab/placebo
Drug: Bevacizumab — Bevacizumab 10mg/kg IV days 1 and 15 of 28 day cycle
  Other Names: Systemic therapy; Avastin
  Arms: paclitaxel/bevacizumab/placebo
Drug: Paclitaxel — Paclitaxel 90mg/m2 1-hour IV infusion Days 1, 8 and 15 of 28 day cycle. Patients will receive standard pre-medication before each paclitaxel treatment to prevent a hypersensitivity reaction.
  Other Names: Systemic therapy; Taxol
  Arms: paclitaxel/bevacizumab/placebo

SUMMARY:
This randomized, double blind, placebo controlled trial will evaluate the impact of adding everolimus to the combination of weekly paclitaxel plus bevacizumab in the first-line treatment of women with HER2-negative metastatic breast cancer. Patients will be randomized (1:1) to receive either paclitaxel/bevacizumab/everolimus (Treatment Arm 1) or paclitaxel/ bevacizumab/placebo (Treatment Arm 2). Patients will be evaluated for response to treatment every 8 weeks; responding and/or stable patients will continue treatment, with re-evaluations every 8 weeks, until tumor progression or

intolerable toxicity occurs. Outcomes will be assessed for each treatment arm

separately. This trial is not intended to compare treatment arms primarily. Any such analyses are exploratory and will be conducted without adjustment for multiple hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients >=18 years of age.
2. Histologically confirmed invasive breast cancer, locally unresectable or metastatic.
3. No prior chemotherapy for MBC. Patients may have received adjuvant or

   neoadjuvant chemotherapy (including taxanes and/or bevacizumab) as long as

   treated was completed >12 months prior to relapse. Prior hormonal therapy in the

   adjuvant or metastatic setting will be permitted.
4. Prior hormonal therapy in the adjuvant or metastatic setting is permitted. Estrogen receptor positive patients should be considered candidates for chemotherapy.
5. HER2-negative breast cancer, defined as follows:

   * FISH-negative (FISH ratio <2.2), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.2).
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Adequate hematologic function, defined by:

   · Absolute neutrophil count (ANC) >1500/mm3
   * Platelet count >=100,000/mm3
   * Hemoglobin >9 g/dL
8. Adequate liver function, defined by:

   · AST and ALT <=2.5 x the upper limit of normal (ULN) or <=5 x ULN in

   presence of liver metastases
   * Total bilirubin <=1.5 x ULN
9. Adequate renal function, defined by:

   · Serum creatinine <=1.5 x ULN or calculated creatinine clearance of

   >=40 ml/min
10. International normalized ratio (INR) <=1.5 or prothrombin time (PT)/partial

    thromboplastin time (PTT) within normal limits (WNL) of the institution (if patient is not on anti-coagulation therapy). Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin are eligible if the INR is stable and within the therapeutic range prior to study treatment initiation.
11. Adequate lipid profile: total cholesterol <=300 mg/dL OR <=7.75 mmol/L and fasting triglyceride 2.5 x ULN. Note: In case one or both of these thresholds are exceeded,the patient can only be included after initiation of appropriate lipid lowering medication.
12. Patients with proteinuria at screening as demonstrated by either:

    · Urine protein creatinine (UPC) ration >1.0 at screening

    or
    * Urine dipstick for proteinuria >=2+ (patients discovered to have

    >=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour

    urine collection and must demonstrate <1 g of protein in 24 hours to be

    eligible).
13. Measurable disease by RECIST criteria.
14. Life expectancy >=12 weeks.
15. Ability to swallow oral medications.
16. Adequate cardiac function, defined by baseline left ventricular ejection fraction (LVEF) value >= normal per institutional guidelines by MUGA scan or

    echocardiogram (ECHO).
17. Adequate recovery from recent surgery.

    * Major surgical procedure >28 days from study entry
    * Minor surgical procedure >7 days from study entry (Portacath placement

    excepted - patients can start treatment <7 days after portacath placement.)
18. Patients with previous history of invasive cancers (including breast cancer) are eligible if definitive treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
19. Patient must be accessible for treatment and follow-up.
20. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

    -

Exclusion Criteria:

1. Patients with active brain metastases or meningeal metastases. Patients who have had brain metastases resected, or have received brain radiation therapy >4 weeks prior to study entry are eligible, if they meet all of the following criteria: 1) residual symptoms < grade 2, 2) no dexamethasone requirement, and 3) follow-up MRI shows regression of lesions after treatment and no new lesions appearing.
2. Previous treatment with an m-TOR inhibitor (sirolimus, temsirolimus, everolimus) or anti-angiogenesis agent unless:

   * in the adjuvant setting, and
   * >=12 months prior to recurrence.
3. Previous radiotherapy for metastatic disease completed <2 weeks prior to study treatment initiation.
4. Patients who are current receiving systemic cancer therapy or have received

   previous systemic therapy within 4 weeks of the start of study drug (e.g.

   chemotherapy, antibody therapy, targeted agents).
5. Women who are pregnant or lactating. All patients with reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug.
6. Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or

   diastolic pressure >100 mmHg, despite optimal medical management.
7. Concurrent use of CYP3A4 inhibitors and inducers from 72 hours prior to initiation of study treatment until the end of treatment with everolimus.
8. Cardiac disease, including: congestive heart failure (CHF) > Class II per New York Heart Association (NYHA) classification; unstable angina (anginal symptoms at rest) or new-onset angina (i.e., began within the last 3 months), or myocardial infarction within the past 6 months; symptomatic CHF, unstable angina pectoris, or cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
9. History of stroke or transient ischemic attack within 6 months prior to first

   bevacizumab dose.
10. Patients with any non-healing wound, ulcer, or long-bone fracture.
11. Patients with clinical history of hemoptysis or hematemesis.
12. Patients with any history of a bleeding diathesis or coagulopathy.
13. Patients with a PEG or G tube cannot be enrolled into this trial.
14. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning bevacizumab.
15. Patients with an impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
16. Patients who have any severe and/or uncontrolled medical conditions or other

    conditions that could affect their participation such as:
    * severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
    * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
17. History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that might affect interpretation of the results of this study, or render the subject at high risk for treatment complications.
18. History of hypersensitivity to Cremophor EL (polyoxyethylated castor oil) or a drug formulated in Cremophor EL, such as paclitaxel.
19. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
20. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
21. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
22. Concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
23. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or its excipients.
24. Patients with a known HIV seropositivity.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (15):
- United States (15):
  - Wilshire Oncology Medical Group, LaVerne, California
  - Eastern Connecticut Hematology Oncology, Norwich, Connecticut
  - Aventura Medical Center, Aventura, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Associates, Bethesda, Maryland
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mid Ohio Oncology/Hematology, Inc./ The Mark H. Zangmeister Center, Columbus, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Fairfax Northern Virginia Hem-Onc, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin/Placebo | Paclitaxel/Carboplatin/Everolimus
Started | 56 (One patient enrolled/randomized but did not start treatment) | 55 (One patient enrolled/randomized but did not start treatment)
Completed | 0 | 0
Not Completed | 56 | 55

BASELINE CHARACTERISTICS:
Population: Includes all enrolled and randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel/Carboplatin/Placebo | Paclitaxel/Carboplatin/Everolimus | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Median (Full Range); unit: Years] | 57 [25 to 79] | 61 [30 to 77] | 58 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival will be measured from Day 1 of study drug administration to disease progression defined by Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 8 weeks until progressive disease, expected average of 18 months
Population: Includes all enrolled and randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Number analyzed (Participants) | 56 | 57
months | 9.1 [6.8 to 10.8] | 7.1 [5.6 to 10.8]

2. Secondary Outcome: Number of Patients With Treatment-related Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: Assessments will be made based on the analysis of reported incidence of treatment-emergent AEs
Time Frame: every 4 weeks until intolerable toxicity occurs
Population: Includes patients who were enrolled, randomized and treated
Measure: Number; unit: participants
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Number analyzed (Participants) | 55 | 56
participants
  Neutropenia | 27 | 26
  Febrile neutropenia | 2 | 2
  Anemia | 23 | 8
  Thrombocytopenia | 12 | 8
  Fatigue | 38 | 29
  Mucositis/stomatitis | 35 | 18
  Neuropathy | 32 | 31
  Diarrhea | 30 | 17
  Rash | 25 | 13
  Nausea/vomiting | 26 | 19
  Epistaxis | 20 | 15
  Arthralgia/myalgia | 19 | 10
  Alopecia | 19 | 27
  Anorexia/weight loss | 18 | 13
  Proteinuria | 17 | 10
  Dysgeusia | 11 | 8
  Headache | 11 | 7
  Hypertension | 10 | 10
  Dyspnea | 10 | 9
  Hypercholesterolemia | 9 | 3

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The number of patients with observed complete response [CR] or partial response [PR]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: every 8 weeks until treatment discontinuation, expected average of 18 months
Population: Includes patients who were enrolled and randomized
Measure: Number; unit: participants
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Number analyzed (Participants) | 56 | 57
participants | 35 | 32

4. Secondary Outcome: Duration of Response (DOR)
Description: Defined as time between date of objective response and date of response to disease progression or death, as defined by RECIST v1.1 criteria. Objective response is defined as either complete response [CR] or partial response [PR]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 8 weeks until treatment discontinuation, expected average 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Number analyzed (Participants) | 35 | 32
months | 7.8 [5.8 to 9.2] | 6.0 [5.2 to 14.5]

5. Secondary Outcome: Overall Survival (OS)
Description: Assessed from Day 1 of study drug administration to date of death due to any cause.
Time Frame: every 8 weeks until treatment discontinuation, expected average 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Number analyzed (Participants) | 56 | 57
months | 17.5 [14.9 to 23.9] | 19.6 [14.0 to 27.2]

ADVERSE EVENTS:
Description: Adverse Event analysis includes only patients who were enrolled, randomized and treated
Arm/Group | Paclitaxel/Bevacizumab/Everolimus | Paclitaxel/Bevacizumab/Placebo
Serious Adverse Events (participants affected / at risk) | 16/55 | 16/56
Other Adverse Events (participants affected / at risk) | 55/55 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Bevacizumab/Everolimus (N=55) | Paclitaxel/Bevacizumab/Placebo (N=56)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (8)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (3) | 2 (3)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CENTRAL LINE INFECTION (Infections and infestations) | 0 (0) | 1 (2)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Bevacizumab/Everolimus (N=55) | Paclitaxel/Bevacizumab/Placebo (N=56)
ANAEMIA (Blood and lymphatic system disorders) | 22 (67) | 8 (25)
LEUKOPENIA (Blood and lymphatic system disorders) | 15 (43) | 10 (23)
NEUTROPENIA (Blood and lymphatic system disorders) | 27 (71) | 24 (57)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 11 (29) | 7 (8)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (10) | 3 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 17 (22) | 17 (26)
DIARRHOEA (Gastrointestinal disorders) | 38 (68) | 24 (37)
DRY MOUTH (Gastrointestinal disorders) | 4 (4) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 5 (6) | 8 (8)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 10 (10)
HAEMORRHOIDS (Gastrointestinal disorders) | 5 (5) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 30 (54) | 25 (34)
ORAL PAIN (Gastrointestinal disorders) | 7 (10) | 1 (3)
STOMATITIS (Gastrointestinal disorders) | 16 (39) | 4 (4)
VOMITING (Gastrointestinal disorders) | 22 (29) | 13 (15)
ASTHENIA (General disorders) | 5 (6) | 7 (7)
FATIGUE (General disorders) | 42 (86) | 37 (76)
MUCOSAL INFLAMMATION (General disorders) | 21 (33) | 14 (21)
OEDEMA PERIPHERAL (General disorders) | 8 (14) | 12 (17)
PAIN (General disorders) | 3 (5) | 5 (6)
PYREXIA (General disorders) | 14 (21) | 7 (9)
SINUSITIS (Infections and infestations) | 11 (19) | 6 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 9 (13)
URINARY TRACT INFECTION (Infections and infestations) | 11 (16) | 12 (15)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (7) | 2 (3)
WEIGHT DECREASED (Investigations) | 16 (24) | 7 (7)
ANOREXIA (Metabolism and nutrition disorders) | 13 (20) | 8 (9)
DEHYDRATION (Metabolism and nutrition disorders) | 8 (8) | 5 (7)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 7 (9) | 3 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 5 (6) | 4 (5)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 (20) | 10 (19)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (11)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (12)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 (13) | 6 (8)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (17) | 7 (8)
DIZZINESS (Nervous system disorders) | 4 (4) | 8 (10)
DYSGEUSIA (Nervous system disorders) | 11 (15) | 9 (11)
HEADACHE (Nervous system disorders) | 19 (24) | 15 (26)
HYPOAESTHESIA (Nervous system disorders) | 3 (3) | 4 (5)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 22 (52) | 27 (52)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 13 (27) | 12 (21)
ANXIETY (Psychiatric disorders) | 6 (9) | 6 (6)
DEPRESSION (Psychiatric disorders) | 8 (10) | 6 (7)
INSOMNIA (Psychiatric disorders) | 10 (10) | 8 (8)
DYSURIA (Renal and urinary disorders) | 1 (2) | 7 (9)
PROTEINURIA (Renal and urinary disorders) | 19 (46) | 12 (24)
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 16 (20)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 13 (18)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 28 (40) | 19 (24)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 6 (7)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (5)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
ALOPECIA (Skin and subcutaneous tissue disorders) | 19 (23) | 30 (38)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 5 (16) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 6 (6) | 14 (20)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
RASH (Skin and subcutaneous tissue disorders) | 22 (36) | 15 (21)
FLUSHING (Vascular disorders) | 2 (2) | 4 (4)
HOT FLUSH (Vascular disorders) | 3 (3) | 8 (10)
HYPERTENSION (Vascular disorders) | 12 (19) | 14 (30)
LYMPHOEDEMA (Vascular disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from the date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish results until 18 mos. after the trial has been completed at all sites.